CLINICAL TRIAL: NCT05601427
Title: A Randomized Controlled Trial Assessing the Efficacy of Surgeon-performed, Intraoperative Adductor Canal Blocks in Same-Day Discharge Total Knee Arthroplasty
Brief Title: Intra-Operative Adductor Canal Blocks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Orthopaedic Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20220573-01H
Record Dates: First submitted 2022-09-20; First posted 2022-11-01 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis; Knee Arthritis; Knee Pain Chronic; Anesthesia
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anesthesiologist-Performed Adductor Canal Block (aACB) (Active Comparator): Patients will get a pre-operative adductor canal block performed by an anesthesiologist.
  Interventions: Procedure: aACB
- Surgeon-Performed Adductor Canal Block (sACB) (Experimental): Patients will get an intra-operative adductor canal block performed by the surgeon
  Interventions: Procedure: sACB

INTERVENTIONS:
Procedure: aACB — The patient will undergo a pre-operative single-shot, ultrasound-guided ACB performed by an anaesthesiologist skilled in regional anaesthesia techniques. The ACB will be performed in a dedicated block room, immediately prior to administration of a spinal anaesthetic.
  Arms: Anesthesiologist-Performed Adductor Canal Block (aACB)
Procedure: sACB — The patient will undergo an intraoperative single-shot ACB performed by the treating surgeon following placement of the TKA components.
  Arms: Surgeon-Performed Adductor Canal Block (sACB)

SUMMARY:
Adductor canal blocks (ACB) have been recommended in total knee arthroplasty (TKA) to provide better control of post-operative pain, facilitate early ambulation, and reduce length of stay in the hospital. ACB is typically done before surgery by an anesthesiologist, which may increase time per case, cost, and requires the specialized skills of an anesthesiologist trained in regional anesthesia. Recent studies have suggested that surgeons can safely and reliably administer the adductor canal blocks (sACB) during surgery. However, there is currently very limited data on the clinical efficacy of such sACBs, and no studies assessing this technique in the context TKA that are discharged the same day. As such, this randomized control trial (RCT) is being done to compare sACBs to conventional anesthesiologist-performed adductor canal blocks (aACB).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 years or older
2. Primary TKA booked as SDD
3. Diagnosis of osteoarthritis

Exclusion Criteria:

1. Inability or refusal to sign informed consent form
2. Non-English or French speaking, and no licensed translator, family member or substitute decision maker available.
3. Non-osteoarthritis primary diagnosis
4. Allergy to analgesic medications
5. Contraindication to spinal and/or regional anaesthesia
6. Any use of opioid pain medication within four weeks of the index procedure(13)
7. Pain catastrophizing scale score ≥16 (8, 9, 14)
8. History of cirrhosis
9. History renal insufficiency
10. History or sensory and/or motor neuropathy to the ipsilateral limb
11. Simultaneous, bilateral TKA
12. Non-TKA prosthesis
13. Scheduled for non-SDD TKA.
14. Preoperative varus/valgus of >10 degrees.
15. Planned General Anaesthetic
16. Use of Intrathecal Morphine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Patient Report Pain | Up to 24 hours
  Mean Numerical Pain Rating Scale (NPRS) scores on discharge
Pain medication use | When spinal anesthesia resolves until 24 hours after surgery
  morphine equivalents of pain medication

SECONDARY OUTCOMES:
Time to discharge | From PACU to discharge
  Post-operative time in minutes to discharge home
Admission to Hospital | Up to 24 hours post-operative
  Failure to discharge home requiring admission
Readmission Rate | Up to 24 hours post-operative
  Number of patients readmitted to the hospital within 24 hours
Timed Up and Go Test | At discharge
  Time is takes, in seconds, to stand, walk 3m, turn around, walk back 3m, and sit back down
Patient Reported Quality of Recovery | At 24 hours post-operative
  Score on the Quality of Recovery-15 questionnaire
Patient Reported Function | pre-operatively, at 2 weeks post-operative
  Difference in scores on the Oxford knee score (questionnaire), rated from 0-48 with 48 being the best functional outcome and 0 being the worst
Patient Reported Quality of Life | pre-operatively, at 2 weeks post-operative
  Difference in scores on the EQ-5D-5L questionnaire (Euro Quality of Life, 5 Dimension, 5 Level), rated from 11111 - 55555, with 11111 being full health and 55555 being worst health
Patient Reported Global Health | pre-operatively, at 2 weeks post-operative
  Difference in scores on the PROMIS-10 - Global Health (questionnaire), which generates T-scores. Higher T-scores indicate better health.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Garceau, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No